CLINICAL TRIAL: NCT06720324
Title: An Open-label Clinical Study on the Efficacy and Safety of CD7-specific CAR-T Cell Injection in the Treatment of CD7-positive Relapsed/Refractory Hematologic Tumors
Brief Title: CD7-specific CAR-T Cell in the Treatment of CD7-positive Relapsed/Refractory Hematologic Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, MEI HENG, : Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7 CAR-T
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Malignancy
Keywords: CD7; CAR-T
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide +CD7-specific CAR-T Cells (Experimental): Patients will received lymphodepletion with fludarabine (30 mg/kg) and cyclophosphamide (300 mg/kg) on day -5, -4, and -3, followed by the infusion of CD7-specific CAR-T Cells with the dose of 1-3×10^6/kg.
  Interventions: Drug: Fludarabine + Cyclophosphamide + CD7-specific CAR-T Cells

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + CD7-specific CAR-T Cells — fludarabine 30 mg/kg on day -5, -4, and -3; cyclophosphamide 300 mg/kg on day -5, -4, and -3; CD7-specific CAR-T Cells on day 0.

SUMMARY:
This study is a single-center, open, prospective single-arm clinical study of patients with CD7 postive relapsed / refractoryhematological tumors to evaluate the safety and efficacy of CD7-specific CAR-T cells in relapsed / refractory hematological tumors while collecting pharmacokinetics and pharmacodynamics indicators of CAR-T cells.

DETAILED DESCRIPTION:
In order to study CD7-targeting CAR-T cell therapy, we constructed a lentiviral CAR structure. The CD7-targeting fragment was cloned into a second-generation CAR structural backbone with 4-1BB and CD3E. Since endogenous CD7 in T cells causes CD7-targeting CAR-T cells to kill each other, we used a natural selection method to prepare CD7-targeting CAR (CD7-CART) T cells that do not express the CD7 protein (CD7-).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of relapsed/refractory hematologic malignancies that meet any of the following criteria:

  1. Recurrence: peripheral blood or bone marrow blasts (proportion>5%) after achieving complete remission after previous standard treatment regimens, or extramedullary disease, including:

     i) Early recurrence within 12 months; ii) Late recurrence of 12 months or more with no remission after one course of standard induction chemotherapy; iii) Relapse after autologous or allogeneic hematopoietic stem cell transplantation.
  2. Refractory: complete remission is not achieved after at least two courses of standard induction therapy, or complete remission is not achieved after first-line or above salvage therapy
* At the time of enrollment screening, bone marrow flow cytometry detected tumor cells as CD7 expression and/or pathological immunohistochemistry of extramedullary lesions was confirmed that tumor cells expressed CD7.
* If tumor cells are detected in peripheral blood during enrollment screening, the immunophenotype of tumor cell surface at the time of flow cytometry detection should be CD4 and CD8 negative. If the surface immunophenotype of peripheral blood tumor cells is not CD4 and CD8 negative, the condition of ≤1% proportion of peripheral blood tumor cells must be met.
* Subjects with the Eastern Cooperative Oncology Group (ECOG) fitness scores of 0 to 2.
* Expected survival over 3 months;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Serum creatinine ≤ 1.5× ULN；
  2. Left ventricular ejection fraction (LVEF) ≥50%;
  3. Baseline peripheral oxygen saturation > 90%;
  4. Total bilirubin ≤ 1.5×ULN; ALT and AST ≤2.5×ULN.
* Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

* Appearance of one of the following cardiac criteria: atrial fibrillation; myocardial infarction in the last 12 months; prolonged QT syndrome or secondary QT extension, as judged by the investigator.

Echocardiography LVSF <30% or LVEF <50%; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV (confirmed by echocardiography within 12 months of treatment).

* Active GVHD.
* History of severe pulmonary function impairment disease.
* Other malignant tumors in the advanced stage.
* Severe infection or persistent infection that cannot be effectively controlled.
* Combined with severe autoimmune disease or innate immune deficiency.
* Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA 500 IU / ml and abnormal liver function] or hepatitis C antibody [HCV-Ab] positive, HCV-RNA above the lower limit of detection of the analytical method and abnormal liver function).
* Human immunodeficiency virus (HIV) infection or syphilis infection.
* History of severe allergies to biological products (including antibiotics).
* Central nervous system disorders, such as uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, etc..
* Female patients are in pregnancy and lactation, or have a pregnancy plan within 12 months.
* Situations where the investigator may increase the risk or interfere with the test results.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) of administering CD7-specific CAR-T Cells In the treatment of relapsed/refractory hematologic tumors | within 3 years after infusion
  Disease overall response rate (ORR) will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Incidence of Treatment-related Adverse Events | Within 3 month after CD19&CD20 CAR-T infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
In vivo expansion and survival of CD7-specific CAR-T Cells in relapsed/refractory hematological malignancies | within 3 years after infusion
  Quantity of CD7 CAR copies in bone marrow, peripheral blood and cerebrospinal fluid will be determined by using flow cytometry and quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Heng, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadelain M, Riviere I, Riddell S. Therapeutic T cell engineering. Nature. 2017 May 24;545(7655):423-431. doi: 10.1038/nature22395. PMID 28541315
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] Turtle CJ, Hanafi LA, Berger C, Gooley TA, Cherian S, Hudecek M, Sommermeyer D, Melville K, Pender B, Budiarto TM, Robinson E, Steevens NN, Chaney C, Soma L, Chen X, Yeung C, Wood B, Li D, Cao J, Heimfeld S, Jensen MC, Riddell SR, Maloney DG. CD19 CAR-T cells of defined CD4+:CD8+ composition in adult B cell ALL patients. J Clin Invest. 2016 Jun 1;126(6):2123-38. doi: 10.1172/JCI85309. Epub 2016 Apr 25. PMID 27111235